

Title: A Phase 1, Open-Label Positron Emission Tomography Study in Healthy Subjects to Determine the Effect of TAK-041 on Amphetamine-Induced Dopamine Release in the CNS After Single-Dose Oral Administration

NCT Number: NCT02959892

SAP Approve Date: 19 May 2017

Certain information within this Statistical Analysis Plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable (PPD) information or company confidential information (CCI).

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.



### STATISTICAL ANALYSIS PLAN

STUDY NUMBER: TAK-041-1002

A Phase 1, Open-Label Positron Emission Tomography Study in Healthy Subjects to Determine the Effect of TAK-041 on Amphetamine-Induced Dopamine Release in the CNS After Single-Dose Oral Administration

Phase 1 TAK-041 Single-Dose PET Study

PHASE 1

Version: Final

**Date:** 19 May 2017

Prepared by:

Based on:

Protocol Version: Amendment 02

Protocol Date: 21 February 2017

#### 1.1 **Approval Signatures**

**Study Title:** 

A Phase 1, Open-Label Positron Emission Tomography Study in Healthy Subjects to Determine the Effect of TAK-041 on Amphetamine-Induced Dopamine Release in the CNS After Single-Dose Oral A.

Administration and subject to the addition of take daily o

| 2.0 | TABLE OF CONTENTS | |
|---|---|---|
| 1.0 | TITLE PAGE | 1 |
| 1. | 1 Approval Signatures | 2 |
| 2.0 | | |
| 3.0 | LIST OF ABBREVIATIONS | 5 |
| 4.0 | OBJECTIVES | 7 |
| 4. | 1 Primary Objective | 7 |
| 4.2 | TABLE OF CONTENTS. LIST OF ABBREVIATIONS OBJECTIVES 1 Primary Objective. 2 Secondary Objective. 3 Additional Objectives. 4 Study Design. 4.4.1 Dose Decisions. ANALYSIS ENDPOINTS. 1 Primary Endpoint. 2 Secondary Endpoint. 3 Exploratory/Additional Endpoints. DETERMINATION OF SAMPLE SIZE. METHODS OF ANALYSIS AND PRESENTATION | 7 |
| 4.3 | 3 Additional Objectives | 7 |
| 4.4 | 4 Study Design | 7 |
| | 4.4.1 Dose Decisions | 10 |
| 5.0 | ANALYSIS ENDPOINTS | 12 |
| 5. | 1 Primary Endpoint | 12 |
| 5.2 | 2 Secondary Endpoint | 12 |
| 5 | 3 Exploratory/Additional Endpoints | 12 |
| 6.0 | DETERMINATION OF SAMPLE SIZE | 13 |
| 7.0 | WETHODS OF THATE I SIS THAT I RESERVITION | |
| 7. | 1 General Principles. | 14 |
| | 7.1.1 Conventions for Missing Data | 14 |
| | 7.1.2 Definition of Study Days and Baseline | |
| | 7.1.3 Derived Datasets and Variables | |
| 7.2 | | |
| 7.3 | 93 | |
| 7.4 | 8 1 | |
| 7.5 | | |
| 7.0 | <b>X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X</b> | |
| 7. | | |
| 7.5 | 8 Efficacy Analysis | |
| 7.6 | Pharmacokinetic/Pharmacodynamic Analysis | |
| 6, | 7.9.1 Pharmacokinetic Analysis | |
| \ | 7.9.2 Pharmacodynamic Analysis | |
| 7. | | |
| 7. | | |
| | 7.11.1 Adverse Events | |
| | 7.11.2 Clinical Laboratory Evaluations | .19 |

| 20 21 22 22 23 23 25 26 26 27 28 28 29 29 20 20 20 20 20 20 21 20 20 20 20 20 21 20 20 20 21 20 20 20 20 21 20 21 20 20 20 20 20 20 21 20 |
|---|
| ons Related to Safety |
| ification of Markedly Abnormal Laboratory Values |
| ormal Changes from Baseline of Vital Signs |
| ormal Changes from Baseline of Vital Signs |
| ormal Changes from Baseline of Vital Signs |
| ification of Markedly Abnormal Orthostatic Changes |
| tedly Abnormal Values for the 12-Lead ECG Parameters27 |
| ightise office |
| Mercial use |

#### 3.0 LIST OF ABBREVIATIONS

%CV [<sup>11</sup>C]PHNO

**ADaM** 

ΑE

ALT

**AMPH** 

aPTT AST

BMI bpm

 $BP_{ND}$ 

**CDISC** 

CI

 $C_{\text{max}}$ 

**CNS CPK** CS

C-SSRS

CV conventional units D2/D3dopamine-2 and -3 **ECG** electrocardiogram

electronic case report form **eCRF** 

ET early termination **GGT** γ-glutamyl transferase

CCI

International Conference on Harmonization

international normalized ratio

MAV MedDRA MRI lower limit of normal lower limit of quantitation not clinically significant markedly abnormal value

Medical Dictionary for Regulatory Activities

magnetic resonance imaging PET positron emission tomography

PHNO (+)-4-propyl-3,4,4a,5,6,10b-hexahydro-2*H*-naphtho[1,2-*b*][1,4]oxazin-9-ol

pharmacokinetics PT preferred term PT prothrombin PTE pretreatment event

To determine brain penetration of single oral doses of TAK-041 and its effects on amphetamine (AMPH)-induced dopamine release in the central nervous system (CNS).

• Hypothesis: at 1 or more dose levels, TAK-041 will per 1

AMPH-induced dopamine rol-

#### 4.2 **Secondary Objective**

To determine a dose/exposure response relationship of TAK-041 on AMPH-induced dopamine release in the CNS.

4.3 **Additional Objectives** 

#### 4.4 **Study Design**

This is a phase 1, open-label clinical study utilizing positron emission tomography (PET) and the radiolabeled dopamine-2 and -3 (D2/D3) receptor agonist PET ligand [11C]-(+)-4-propyl-3,4,4a,5,6,10b-hexahydro-2H-naphtho [1,2-b][1,4]oxazin-9-ol ( $[^{11}C]$ PHNO) to evaluate the effects of single oral doses of TAK-041 on AMPH-induced dopamine release in the brain in 12 healthy male subjects.

Subjects will continue to be enrolled until 12 evaluable subjects complete all procedures. Each subject will have 1 magnetic resonance imaging (MRI) brain scan and 3 [11C]PHNO PET scans. The MRI brain scan will be performed for all subjects without gadolinium contrast and will be interpreted at the during the Screening Period to determine eligibility. The results of this MRI brain scan will also be used during the study to delineate the anatomical regions of interest for individual PET images.

The study consists of 2 Confinement Periods for each subject during which the PET scans will occur at the . Confinement Periods 1 and 2 will be separated by an interval of 5 to 45 days.

## Confinement Period 1:

The first [11C]PHNO PET scan occurs on Day 1 to serve as the Baseline scan to determine the nondisplaceable binding potential (BP<sub>ND</sub>) in striatum under untreated conditions for each subject.

On Day 2, the subject will receive a single oral 0.5 mg/kg dose of AMPH, followed by a [<sup>11</sup>C]PHNO PET scan at approximately 3 hours post-AMPH dose in order to establish BP<sub>ND</sub> in striatum after AMPH-induced dopamine release as compared to Baseline.

### • Confinement Period 2:

On Day 1, the subject will receive a single oral dose of TAK-041 up to 40 mg, followed by a single oral 0.5 mg/kg dose of AMPH approximately 2 hours after the dose of TAK-041, followed by a [<sup>11</sup>C]PHNO PET scan at approximately 3 hours post-AMPH administration.

Blood samples for pharmacokinetic (PK) analysis of AMPH will be collected prior to AMPH administration, 1 and 2 hours post-AMPH administration, and immediately prior to and after the [ $^{11}$ C]PHNO PET scan to measure plasma levels of AMPH. PK blood samples will be collected 1, 2, 12, and 24 hours after TAK-041 administration, immediately prior to and after the [ $^{11}$ C]PHNO PET scan, and during each Follow-up Visit. Following discharge from Confinement Period 2, subjects will return to the site for PK and safety assessments after  $7 \pm 2$  days, and then return for approximately 3 Follow-up Visits (once every 4 weeks) or until the concentration of TAK-041 in plasma is <5% of the subject's maximum observed plasma concentration ( $C_{max}$ ).

Amphetamine tablets will be provided as the commercial product dexamfetamine sulphate [1] with the manufacturer's original label, and will be sourced locally by the study site. Using data from the TAK-041-1001 study, AMPH will be administered at the approximate time to reach  $C_{max}$  (t<sub>max</sub>) (plasma) of TAK-041 to allow an informative evaluation of TAK-041 coadministered with amphetamine. The [ $^{11}$ C]PHNO PET scan will start at the approximate t<sub>max</sub> (plasma) of AMPH (estimated to be 3 hours post-AMPH dose). The starting dose of TAK-041 in this study will be 20 mg, a dose that has been demonstrated to be well-tolerated in the TAK-041-1001 study and has achieved exposures indicative of the predicted pharmacologically active exposures of TAK-041. A single dose level of 40 mg TAK-041 has also been shown to be well-tolerated in the TAK-041-1001 study and may be evaluated in this study to explore the exposure-response relationship of TAK-041. The highest dose of AMPH that will be administered will be an oral dose of 0.5 mg/kg. This dose has been demonstrated to be safe and well-tolerated in healthy subjects and is a dose which has been shown to induce dopamine release in AMPH-challenge studies [2, 3].

Safety and tolerability will be assessed through all study visits, including collecting blood and urine samples for laboratory tests. Subjects will complete scheduled study assessments according to the Schedule of Study Procedures in the protocol [4].

| Statistical Allalysis 1 la | 111 |
|----------------------------|-----|
| JCI | |

Each subject will report to on approximately 8 occasions:

- 1. Screening Visit to determine eligibility (-28 to -2 days prior to Confinement Period 1/Day 1): The Screening brain MRI may be performed on a day separate from the other screening procedures, and will be performed and interpreted at the other screening activities have been performed and results assessed. MRI should be performed early enough so that MRI scan results are available prior to Baseline Imaging for Confinement Period 1.
- 2. Confinement Period 1 (Day -1 to Day 3): admission to CCI (Day -1), 1 day prior to Baseline [11C]PHNO PET imaging on Day 1; AMPH administration and postdose [11C]PHNO PET imaging on Day 2; discharge on Day 3, the day following the postdose [11C]PHNO PET imaging. All subjects will undergo a single predose [11C]PHNO PET scan on Day 1 and a single postdose [11C]PHNO PET scan on Day 2.
- 3. Confinement Period 2 (5 to 45 days after discharge from Confinement Period 1): admission to Color (Day -1) 1 day prior to TAK-041 and AMPH administration and postdose [11C]PHNO PET imaging (Day 1), discharge on Day 2, the day following the postdose [11C]PHNO PET imaging. All subjects will undergo a single postdose [11C]PHNO PET scan on Day 1 of Confinement Period 2.
- 4. Follow-up Safety and PK Assessment Visits (Days 8-92): Following discharge from Confinement Period 2, subjects will return to the site for PK and safety assessments after 7±2 days, and then return for approximately 3 Follow-up safety and PK assessment Visits (once every 4 weeks) or until the concentration of TAK-041 in plasma is <5% of the subject's C<sub>max</sub> (see Section 9.3.2 in the protocol [4]).
- 5. Study Exit/Final Visit: At the end of each Follow-up Visit, the next visit will be scheduled approximately 4 weeks later. If, when the PK results are available, the subject's plasma PK concentration value was <5% of their C<sub>max</sub> value, the site and subject will be informed that their next scheduled visit will be considered their Study Exit/Final Visit (see Section 9.3.3 in the protocol [4]). Subjects who prematurely discontinue the study will have the same assessments for Study Exit/Final Visit performed on their last day in the study, if possible.

A schematic of the study design is shown in Figure 4.a.

Plogistical limitations (such as tracer synthesis failure) prevent a Baseline PET scan from being performed at the scheduled time point, the Confinement Period may be extended or cut short and rescheduled. If a postdose PET scan is delayed, it may be necessary to end the Confinement Period early and reschedule after a sufficient interval.

CCL

The date the final subject completes the Follow-up Call/Visit will be considered the end of study date for transparency reporting.

Figure 4.a Schematic of Study Design

| Screening | | Confinem | ent Period | 1 | Interval (a) | Con | ifinement Po | eriod 2 | Follow-up<br>Visits (b) | Study<br>Exit/Final<br>Visit<br>ET(c) |
|---|---|---|---|---|---|---|---|---|---|---|
| Days -28 to -2 | Day -1 | Day 1 | Day 2 | Day 3 | 5-45 days | Day -1 | Day 1 | Day 2 | Days 8-92<br>(±2) | |
| CCI | Check-in | PET<br>Imaging<br>Baseline | АМРН | CCI<br>Discharge | | Check-in | FAK-041+<br>AMPH | CCI<br>Discharge | Return to CCI for safety and PK assessments | Return to for safety assessments |
| | | | PET<br>Imaging<br>postdose | | | Asilie | PET<br>Imaging<br>postdose | | | |

ET=early termination

Note: Subjects who drop out prior to completion of all PET scans will have assessments done as described in Section 9.3.3 of the protocol [4] for ET and a follow-up telephone call approximately 2 days after the ET Visit.

- (a) There will be a 5 to 45 day interval between confinement periods beginning after discharge from Confinement Period 1.
- (b) Following discharge from Confinement Period 2, subjects will return to the site for PK and safety assessments after  $7 \pm 2$  days, and then return for approximately 3 Follow-up PK and safety assessment Visits (once every 4 weeks) or until the concentration of TAK-041 in plasma is <5% of the subject's  $C_{max}$ .
- (c) At the end of each Follow-up Visit, the next visit will be scheduled approximately 4 weeks later. If, when the PK results are available, the subject's PK was <5% of their  $C_{max}$  value, the site and subject will be informed that their next scheduled visit will be considered their Study Exit/Final Visit.

### 4.4.1 Dose Decisions

All decisions concerning dose levels will be made by the sponsor and the CCI

This study will utilize an adaptive design to determine the dose(s) of AMPH and TAK-041 to be administered:

- The first 4 subjects in this study will receive a 20 mg dose of TAK-041 and a 0.5 mg/kg dose of AMPH.
- If the results from these subjects do not show at least 10% blunting (lower bound of the one-sided 95% confidence interval [CI]  $\leq$ 10%) in the AMPH-induced dopamine release in the striatum (as measured by changes in BP<sub>ND</sub>), the next 4 subjects will receive a 40 mg dose of TAK-041, and a 0.5 mg/kg dose of AMPH.

- erms of Use If the results from the first 4 subjects show 10% or more blunting (lower bound of the onesided 95% CI > 10%) in the AMPH-induced dopamine release in the striatum (as measured by changes in BP<sub>ND</sub>), the next 4 subjects will receive a 5 mg dose of TAK-041 (based on observed exposures in the TAK-041-1001 study) and a 0.5 mg/kg dose of AMPH.
- Depending on the results from the first 8 subjects, the last 4 subjects may receive either:
  - A dose of TAK-041 between 5 and 40 mg (based on exposures evaluated in the TAK-041-1001 study) and a 0.5 mg/kg dose of AMPH (if both previously tested TAK-041 dose levels showed a blunting of AMPH-induced dopamine release); or
  - A 40 mg dose of TAK-041 and a 0.25 mg/kg dose of AMPH.

Decisions regarding the doses of TAK-041 and AMPH that Subjects 5 to 12 will receive will be based on discussions between Takeda and the The dose range for TAK-041 is limited by exposures observed in the TAK-041-1001 study. Previous studies with property of Takeda. For non-commercial use only and party of Takeda. For non-commercial use only and party of Takeda. AMPH used doses ranging from 0.3 to 0.5 mg/kg. Testing with the lower AMPH dose is driven by considerations to avoid overstimulation of the dopamine system.

### 5.0 ANALYSIS ENDPOINTS

## 5.1 Primary Endpoint

• The change in BP<sub>ND</sub> in the TAK-041+AMPH condition compared to AMPH alone.

The primary endpoint will be collected, analyzed, and processed by an outside vendor. No analyses are planned on these measures as part of this statistical analysis plan (SAP).

## 5.2 Secondary Endpoint

• The change in BP<sub>ND</sub> in the TAK-041+AMPH condition compared to AMPH alone as a function of the dose of TAK-041 administered.

The secondary endpoint will be collected, analyzed, and processed by an outside vendor. No analyses are planned on these measures as part of this SAP.



Using previously reported data [5], and assuming a 16% standard deviation for the relative change in BP<sub>ND</sub> for high uptake regions of interest, 12 subjects will provide approximately 80% power to detect a 20% relative change in BP<sub>ND</sub> when values from the TAK-041+AMPH condition are compared to AMPH alone condition using a 2-sample 2-sided t-test with 0.05 significance level. The power for the other regions of interest will be more than 80%. enterly st with 0.05' an 80%. July and subject to the adopticable only adopticable only adoptic

This SAP was developed based on International Conference on Harmonization (ICH) E3 and E9 Guidelines. This SAP should be read in conjunction with the study protocol and electronic report forms (eCRF). This version of the SAP was developed using the Protocol TAK-041-1002, amendment 02 day.

All study-related raw data, including derived data, will be presented in data listings. Continuous data will be summarized using: number of subjects (N), mean, standard deviation (SD), median, minimum, and maximum, where appropriate. Categorical data will be summarized using the number and percentage of subjects for each category where appropriate.

Arithmetic means, geometric means, and medians will be presented to more decimal place than the recorded data. SDs will be presented to 2 more decimal places than the recorded data.

PET, MRI, and wearable device data collected on the eCRF will be included in listings. PET, MRI, and wearable device data collected by outside vendors will not be listed. All other study related raw and derived data for enrolled subjects will be presented in listings.

All data analyses will be generated using SAS System® Version 9.2 or higher.

# 7.1.1 Conventions for Missing Data

There will be no imputation of incomplete or missing data. Decisions regarding inclusion or exclusion of data from an analysis for subjects who are noncompliant with the dose schedule, or who have incomplete data, will be made on a case-by-case basis, but the data will be presented in data listings regardless.

Plasma concentrations that are below the lower limit of quantitation (LLOQ) will be treated as zero in the summarizing of concentration values and deriving of PK parameters. These values will be flagged in the data listings, and deviations from this convention may be considered on a case-by-case basis as deemed appropriate.

# 7.1.2 Definition of Study Days and Baseline

Study Day bis defined as the date of the first dose of [11C]PHNO PET tracer. Study days prior to the first dose of [11C]PHNO will be calculated as: {date of assessment/event - date of first dose of [11C]PHNO}. Study days on or after the first dose of [11C]PHNO will be calculated as: {date of assessment/event - date of first dose of  $[^{11}C]PHNO + 1$ .

Day within a period is relative to the date of first dose of study drug ([11C]PHNO, AMPH, or TAK-041) in each confinement period.

Study baseline is defined as the last observed value prior to the first administration of study drug ([11C]PHNO, AMPH, or TAK-041).

### 7.1.3 Derived Datasets and Variables

Derived datasets will be generated according to Clinical Data Interchange Standards Consortium (CDISC) guidance documents: Analysis Data Model (ADaM) Implementation Guide, Version 1.0 or higher.

The following analysis sets will be used for analysis and presentation of the study data:

Safety Set

The safety set will consist of all subjects who are enrolled and receive a dose of study drug ([11C]PHNO, AMPH, or TAK-041) as part of this study. Subjects in this analysis set will be used for demographic, baseline characteristics, and safety summaries.

Pharmacokinetic Set

The PK set will consist of all subjects who receive either AMPH or TAK-041 and have at least 1 measurable plasma concentration for AMPH or TAK-041

#### 7.3 **Disposition of Subjects**

Disposition of all screened subjects will be tabulated (count and percent); there will be no inferential analysis of subject disposition data.

Disposition of screen failure subjects including the primary reasons for failure (i.e., pretreatment event (PTE)/AE, significant protocol deviation, lost to follow-up, voluntary withdrawal, study termination, did not meet entrance criteria, or other) will be presented in a data listing.

Disposition of all enrolled subjects will be tabulated by TAK-041+AMPH dose combination and overall. Categories will include.

- All subjects dosed (denominator).
- Subjects who were enrolled but not dosed, if applicable.
- Subjects who completed all study drugs.
- Subjects who prematurely discontinued study drugs.
- Subjects who completed all study visits.
- Subjects who prematurely discontinued study visits.

Primary reasons for discontinuation of study drugs and/or study visits, as entered on the eCRF, will be tabulated. Reasons for discontinuation include PTE/AE, significant protocol deviation, lost to follow-up, voluntary withdrawal, study termination, and other.

Disposition information for enrolled subjects, including study drug dose level, date of first dose of study drug, date and study day of last dose of study drug, date and study day of last visit, and reason for premature discontinuation of study drugs/study visits (if applicable), will be listed. A

reins of Use listing of inclusion/exclusion criteria not met will be provided for enrolled subjects who did not meet at least one entrance criterion.

Significant protocol deviations captured on the eCRF will be listed.

#### 7.4 **Demographic and Other Baseline Characteristics**

Demographic data will be summarized by assigned TAK-041+AMPH dose combination and overall. Descriptive statistics (N, mean, SD, median, minimum, and maximum) will be generated for continuous demographic variables and baseline characteristics variables (e.g., age at informed consent, height (cm) at screening, weight (kg) at baseline, and body mass index (BMI, kg/m<sup>2</sup>) at screening). The number and percentage of subjects in each class of the categorical demographic variables and baseline characteristics variables (e.g., gender, race, smoking history, alcohol history, and caffeine consumption) will also be tabulated. Individual subject demographic and baseline characteristics data will be listed by site and subject number.

Individual demographic characteristics, date of informed consent, and reason for screen failure will be listed for subjects who are screened but not enrolled in the study.

Race will be recorded on the eCRF as American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or Other Pacific Islander, and White. Subjects who identify themselves as belonging to more than 1 race on the eCRF will be classified as multiracial for summaries and each race selected will be listed.

There will be no inferential analysis of demographic and baseline characteristics.

#### **Medical History and Concurrent Medical Conditions** 7.5

Medical history is defined as significant conditions or diseases relevant to the disease under study that stopped at or prior to signing of informed consent. Concurrent medical conditions are defined as significant conditions or diseases ongoing or present at signing of informed consent.

Medical history and concurrent medical conditions will be coded using the Medical Dictionary for Drug Regulatory Activities (MedDRA, version 19 or higher) coding system.

All medical history and concurrent medical condition data will be listed by site and subject number. The listing will contain subject identifier, study drug dose level, system organ class (SOC), preferred term (PT), and a detail of the medical history or concurrent condition.

There will be no inferential analysis of medical history and concurrent medical conditions.

# **Medication History and Concomitant Medications**

Medication history information includes any medication relevant to eligibility criteria stopped at or within 30 days prior to signing of informed consent. Concomitant medications include any medications, other than study drug, taken at any time between informed consent and the end of the study.

Medication history and concomitant medications will be coded using the World Health Organization Drug Dictionary (WHOD h 2016 Enhanced or higher. All medication history and concomitant medications will be listed by site and subject number. The listings will contain subject identifier, study drug dose level, WHODrug preferred medication name, dose, unit, frequency, route, start date, stop date, whether the medication was ongoing, and reason for use.

There will be no inferential analysis of medication history and concomitant medications.

#### 7.7 **Study Drug Exposure and Compliance**

The date and time of each study drug ([11C]PHNO, AMPH, or TAK-041) for each subject will be reported in the data listing. Listings and descriptive statistics of PK plasma concentrations for AMPH and TAK-041 will be provided for all subjects. No other summary statistics for the extent of exposure to study drug or compliance calculations will be performed for this study.

## 7.8

Not applicable.

## 7.9

Pharmacokinetic/Pharmacodynamic Analysis
Pharmacokinetic Analysis
lood samples for 3 Serial blood samples for determination of AMPH and TAK-041 will be collected according to Figure 7.a.

Figure 7.a Collection of Blood Samples for Pharmacokinetic Analysis

| Analyte | Matrix | Period | Scheduled Time (hours) |
|---|---|---|---|
| AMPH | Plasma | 1 and 2 | Predose (within 60 minutes prior to dosing), 1 and 2 hours post-AMPH administration, and immediately prior to and after [11C]PHNO PET scan. |
| TAK-041 | Plasma | 201 | 1, 2, 12, and 24 hours post-TAK-041 administration, immediately prior to and after the [11C]PHNO PET scan, and during each Follow-up Visit. |

Blood samples for TAK-041 PK will also be collected at ET if TAK-041 has been administered. All PK summaries and analyses will be based on the PK set.

Concentrations of AMPH and TAK-041 in plasma will be summarized by dose level over each scheduled sampling time point using descriptive statistics (n, arithmetic mean, SD, %CV, median, minimum, and maximum). Individual plasma concentration data versus time will be presented in a data listing.

Plasma concentrations that are below the LLOQ will be treated as zero in the summarization of concentration values. These values will be flagged in the data listings and deviations from this convention may be considered on a case-by-case basis as deemed appropriate.

The need of using the plasma concentrations collected from this study in a PK analysis will be evaluated. If deemed appropriate, a PK analysis plan will be prepared and address the planned analysis.

## 7.9.2 Pharmacodynamic Analysis

Not applicable.

#### 7.10 Other Outcomes

PET, MRI, and wearable device data collected on the eCRF will be included in listings.

The imaging analysis (PET and MRI) will be conducted by an outside vendor and are not included in this SAP.



### 7.11 Safety Analysis

The safety endpoints including AEs, clinical laboratory parameters, vital sign parameters, 12-lead ECG parameters will be summarized and described in data listings. The Safety Set will be used for all summaries of safety parameters. Physical examination and C-SSRS will be described in data listings.

### 7.11.1 Adverse Events

A treatment-emergent adverse event (TEAE) is defined as an AE or a serious AE that occurs or gets worse after receiving the first study drug ([11]C]PHNO, AMPH, or TAK-041) and until Study Exit/Final Visit. A PTE is defined as any untoward medical occurrence occurs prior to first study drug ([11]C]PHNO, AMPH, or TAK-041).

PTE and TEAE verbatim reported terms will be coded by SOC and PT using MedDRA (version 19 or higher) coding system.

TEAEs will be listed and included in the summary tables. TEAEs will be summarized by assigned TAK-041+AMPH dose combination and overall. For each TAK-041+AMPH dose combination, TEAE will be summarized by [\begin{subarray}{c} \begin{subarray}{c} \text{I} \cdot \end{subarray} \text{PHNO Alone (Period 1 Day 1 after the dosing of [\begin{subarray}{c} \begin{subarray}{c} \text{I} \cdot \end{subarray} \text{PHNO tracer and before the dosing of AMPH on Day 2 of Period 1), AMPH Alone (Period 1 Day 2 after the dosing of AMPH and before the dosing of the tracer), AMPH+[\begin{subarray}{c} \begin{subarray}{c} \text{I} \cdot \end{subarray} \text{PINO (after the tracer administration on Day 2 of Period 2 Day 1 after the TAK-041 dosing and before the dosing of AMPH), TAK-041 Alone (Period 2 Day 1 after the dosing of AMPH and before the dosing of tracer), and TAK-041+AMPH+[\begin{subarray}{c} \begin{subarray}{c} \begin{subarray}{c} \text{I} \end{subarray} \text{PINO (Period 2 Day 1 after the tracer administration to Study Exit/Final Visit) according to time of onset, and the Entire Study (after the first dose of study drug and until Study Exit/Final Visit).

In general, TEAEs will be tabulated at the following levels: overall summary (subjects with at least 1 AE), by the MedDRA SOC and the MedDRA PT. The tables will include the number and percentage (N [%]) of subjects. The following summary tables will be generated:

- Overview of Treatment-Emergent Adverse Events.
- Treatment-Emergent Adverse Eve

- Treatment-Emergent Adverse Events by Preferred Term, sorted by the frequency of the overall summary from the most to the least.
- Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term.
- Relationship of Treatment-Emergent Adverse Events to Study Drug by System Organ Class and Preferred Term.
- Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term.
- Intensity of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- Intensity of Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term.

In addition, subject mappings for the TEAEs by SOC and PT will be generated.

When calculating the frequency and percentage of subjects who reported TEAEs, a subject will be counted only once for each SOC or PT when multiple TEAEs are coded to the same SOC or PT. For the intensity or relatedness summaries, if a subject reports multiple TEAEs coded to the same SOC or PT, the TEAE with maximum intensity or strongest relationship will be included in the summary.

For TEAE summaries by treatment interval ([41C]PHNO Alone, AMPH Alone, AMPH+[11C]PHNO, TAK-041 Alone, TAK-041+AMPH, and TAK-041+AMPH+[11C]PHNO), subjects reporting more than one occurrence within a treatment interval for the term (level) being summarized will be counted only once for that interval using the most extreme incident (most severe for the severity tables and related for the relationship to study drug tables). For summaries by Entire Study, subjects reporting more than one occurrence during the Entire Study for the term (level) being summarized will be counted only once using the most extreme incident (most severe for the severity tables and related for the relationship to study drug tables).

AEs with missing intensity will be listed as such in the AE listings, however, will be summarized as severe in summary tables. If the relationship of an event is missing, the relationship for the event will be considered to have been related.

Data listings will be provided for TEAEs and PTEs.

## 7.11.2 Clinical Laboratory Evaluations

Clinical safety laboratory tests include hematology, chemistry, urinalysis, and diagnostic screening. Please refer to Table 9.b in the protocol [4] for a list of all clinical laboratory tests.

All laboratory test parameters will be displayed in individual subject data listings in both International System of Units (SI) and conventional units (CV). For test results not in SI units, the conversion to SI units will be done in derived analysis data sets using the known conversion

factors. All summaries and analyses will be based on the values using SI units unless otherwise stated.

Descriptive statistics (N, mean, SD, median, minimum, and maximum) of clinical laboratory tests for baseline, post-baseline, and change from baseline to each post-baseline visit will be presented by assigned TAK-041+AMPH dose combination and overall for Confinement Period 1 and Confinement Period 2 through Study Exit. Baseline is defined as the last observed value prior to the first administration of study drug ([11C]PHNO, AMPH, or TAK-041). Unscheduled laboratory assessments will be excluded from the summary statistics unless it is for the baseline derivation. Note that urinalysis tests with character results, such as protein and nitrite, will only be listed. No inferential statistics will be presented.

Individual results for hematology and chemistry laboratory tests that meet the Takeda predefined laboratory markedly abnormal value (MAV) criteria in Appendix A will be indicated in the data listing. If a subject has a MAV for a particular laboratory test, all visits for that subject for that parameter will be listed. The number and percentage of subjects with at least 1 post-baseline markedly abnormal laboratory test result will be summarized by TAK-041+AMPH dose combination and overall. The mapping of the subjects who meet the MAV criteria will be listed as a table by TAK-041+AMPH dose combination and overall. All observations, including ones at unscheduled visits, will be included in the MAV mapping and summaries.

All clinical laboratory data will be listed. The listing will include site number, subject identifier, age (at informed consent), gender, study drug dose level, study visit, and sample collection date. Laboratory data outside of the normal reference range will be indicated in the data listing. In addition, MAVs will be flagged.

## 7.11.3 Vital Signs

Vital sign parameters include oral body temperature, blood pressure, respiratory rate, pulse, and weight. Pulse and blood pressure will be measured after 5 minutes supine. Orthostatic pulse and blood pressure will be measured after standing for 2 minutes. Please refer to Table 9.a in the protocol [4] for schedules of vital sign assessments.

Descriptive statistics (N, mean, SD, median, minimum, and maximum) of vital sign parameters for baseline, post-baseline, and change from baseline to each post-baseline visit will be summarized by TAK-041+AMPH dose combination and overall by scheduled time point. Baseline is defined as the last observed value prior to the first administration of study drug ([11C]PHNO, AMPH, or TAK-041). Unscheduled vital sign assessments will be excluded from the summary statistics unless it is for the baseline derivation. No inferential statistics will be presented.

Individual results for vital sign measurements that meet the Takeda predefined vital signs MAV criteria in Appendix B will be indicated in the data listing. If a subject has a MAV for a particular vital sign parameter, all visits for that subject for that parameter will be listed. The number and percentage of subjects with at least 1 post-baseline markedly abnormal vital sign measurement will be summarized by TAK-041+AMPH dose combination and overall. The mapping of the subjects who meet the listed as a table by TAK-

041+AMPH dose combination and overall. All observations, including ones at unscheduled visits, will be included in the MAV mapping and summaries.

ns of Use Orthostatic hypotension, identified by the criteria defined in Appendix C, will be calculated at every time point where standing and supine measurements are available using the formula: standing vital measurement - supine vital measurement. The mapping of the subjects who meet the criteria for orthostatic hypotension will be listed as a table by TAK-041+AMPH dose combination and overall. All orthostatic hypotension observations, including ones at unscheduled visits, will be included in the subject mapping.

All vital sign data will be presented in the data listing. The listing will include site number, subject identifier, age (at informed consent), gender, study drug dose level, study visit, and sample collection date. Vital sign MAVs will be flagged.

### 7.11.4 12-Lead ECGs

ECG parameters include heart rate, PR interval, RR interval, QR interval, QT interval, QT interval corrected with the Bazett correction method (QTcB), and QT interval corrected with the Fridericia correction method (QTcF). Please refer to Table 9.c in the protocol [4] for schedules of ECG assessments.

Descriptive statistics (N, mean, SD, median, minimum, and maximum) of ECG parameters for baseline, post-baseline, and change from each baseline to each post-baseline visit will be summarized by TAK-041+AMPH dose combination and overall by scheduled time point. Baseline is defined as the last observed value prior to the first administration of study drug ([11C]PHNO, AMPH, or TAK-041). Only the scheduled measurements will be included in the summary unless it is for the baseline derivation. No inferential statistics will be presented.

Individual results for 12-lead ECG measurements that meet the Takeda predefined 12-lead ECG MAV criteria in Appendix D will be indicated in the data listing. If a subject has a MAV for a particular ECG parameter all visits for that subject for that parameter will be listed. The number and percentage of subjects with at least 1 post-baseline markedly abnormal 12-lead ECG measurement will be summarized by TAK-041+AMPH dose combination and overall. The mapping of the subjects who meet the MAV criteria will be listed as a table by TAK-041+AMPH dose combination and overall. All observations, including ones at unscheduled visits, will be included in the MAV mapping and summaries.

Overall ECG interpretation category (within normal limits, abnormal not clinically significant [NCS], abnormal clinically significant [CS]) is collected in the eCRF at each scheduled visit. Shifts in ECG interpretation will be presented as cross-tabulations (baseline versus each postbaseline visit) of numbers of subjects with normal, abnormal NCS, and abnormal CS interpretations with missing, if applicable, and total categories by TAK-041+AMPH dose combination and overall by scheduled time point. Baseline is defined as the last observed value prior to the first administration of study drug ([11C]PHNO, AMPH, or TAK-041). Unscheduled ECG assessments will be excluded unless it is for the baseline derivation.

reins of Use All ECG data will be presented in the data listing. The listing will include site number, subject identifier, age (at informed consent), gender, study drug dose level, study visit, and sample collection date. ECG MAVs will be flagged.

## 7.11.5 Other Observations Related to Safety

the application there applies the second Physical examination findings and C-SSRS will be presented in data listings. No summary tables will be provided.

#### 7.12 **Interim Analysis**

No formal interim analysis is planned.

#### **Changes in the Statistical Analysis Plan** 7.13

Aiffer from and gulpies only and gulpies on gulpie Analyses described in the statistical analysis plan do not differ from those specified in the

### 8.0 REFERENCES

- 1. Dexamfetamine sulphate 5 mg tablets. Summary of Product Characteristics. Middlesex, UK: Auden Mckenzie (Pharma Division) Ltd, Revised 16 November 2015.
- 2. Abi-Dargham A, Gil R, Krystal J, Baldwin RM, Seibyl JP, Bowers M, et al. Increased striata dopamine transmission in schizophrenia: confirmation in a second cohort. Am J Psychiatry 1998;155(6):761-7.
- 3. Weidner LD, Paris A, Frankle WG, Narendran R. Safety of oral amphetamine administered during positron emission tomography scans in medically screened humans. PLoS One 2015;10(12):e0140647.
- 4. A Phase 1, Open-Label Positron Emission Tomography Study in Healthy Subjects to Determine the Effect of TAK-041 on Amphetamine-Induced Dopamine Release in the CNS After Single-Dose Oral Administration. Takeda Development Center Europe, Ltd., Protocol No. TAK-041-1002, Amendment 02, dated 21 February, 2017.
- 5. Shotbolt P, Tziortzi AC, Searle GE, Colasanti A, van der Aart J, Abanades S, et al. Within-Jod Flow of Takeda. For non-commercial use only subject comparison of [11C]-(+)-PHNO and [11C]raclopride sensitivity to acute amphetamine challenge in healthy humans. J Cereb Blood Flow Metab 2012;32(1):127-36.

# Appendix A Criteria for Identification of Markedly Abnormal Laboratory Values

## Hematology—Criteria for Markedly Abnormal Values

| Parameter | Unit | Low Abnormal | High Abnormal |
|---|---|---|---|
| Hemoglobin | Both | <0.8 × LLN | >1.2 × ULN |
| Hematocrit | Both | <0.8 × LLN | >1.2 × ULN |
| RBC count | Both | <0.8 × LLN | >1.2 × ULN |
| WBC count | Both | <0.5 x LLN | >1.5 x ULN |
| Platelet count | Conventional | $<75 \times 10^3/\mu L$ | $>600 \times 10^3/\mu L$ |
| | SI | <75 x 109/L | >600 x 109/L |
| PT/INR | Both | | >1.5 × ULN |
| aPTT | Both | | >1.5 × ULN |

aPTT= activated prothrombin time, INR=international normalized ratio, LLN=lower limit of normal, RBC=red blood cell, ULN=upper limit of normal, WBC=white blood cell, PT=prothrombin.

# Serum Chemistry—Criteria for Markedly Abnormal Values

| | | 5 | |
|----------------------|--------------|--------------|---------------|
| Parameter | Unit | Low Abnormal | High Abnormal |
| ALT | Both | | >3x ULN |
| AST | Both | | >3x ULN |
| GGT | Both | (1) | >3x ULN |
| Alkaline phosphatase | Both | 0 | >3x ULN |
| Chloride | Conventional | <75 mEq/L | >126 mEq/L |
| | SI | <75 mmol/L | >126 mmol/L |
| Total bilirubin | Conventional | | >2.0 mg/dL |
| | SI | | >34.2 μmol/L |
| Direct bilirubin | Both | | >2 ULN |
| Albumin | Conventional | <2.5 g/dL | |
| | SI | <25 g/L | |
| Total protein | Both | <0.8x LLN | >1.2x ULN |
| Creatinine | Conventional | | >2.0 mg/dL |
| | SI | | >177 μmol/L |
| Blood urea nitrogen | Conventional | | >30 mg/dL |
| | SI | | >10.7 mmol/L |
| Sodium | Conventional | <130 mEq/L | >150 mEq/L |
| . * | SI | <130 mmol/L | >150 mmol/L |
| Potassium ** | Conventional | <3.0 mEq/L | >6.0 mEq/L |
| CO | SI | <3.0 mmol/L | >6.0 mmol/L |
| CPK | Both | | >5x ULN |
| Glucose | Conventional | < 50 mg/dL | >350 mg/dL |
| × ` | SI | < 2.8 mmol/L | >19.4 mmol/L |
| Creatine kinase | Conventional | | >5 × ULN |
| | SI | | >5 × ULN |
| Bicarbonate | Conventional | <8.0 mEq/L | |
| | SI | <8.0 mmol/L | |
| Calcium | Conventional | <7.0 mg/dL | >11.5 mg/dL |
| | SI | <1.75 mmol/L | >2.88 mmol/L |

ALT=alanine aminotransferase, AST=aspartate aminotransferase, CPK=creatine phosphokinase, GGT= $\gamma$ -glutamyl transferase, LLN=lower limit of normal, ULN

# Appendix B Criteria for Abnormal Changes from Baseline of Vital Signs

| Parameter | Unit | Lower Criteria | Upper Criteria | 7/1 |
|---|---|---|---|---|
| Pulse | bpm | <50 | >120 | 10, |
| Systolic blood pressure | mm Hg | <85 | >180 | 0 |
| Diastolic blood pressure | mm Hg | <50 | >110 | |
| Body temperature | °C | <35.6 | >37.7 | |
| Parameter Pulse Systolic blood pressure Diastolic blood pressure Body temperature | n.commercial use | only and subject | to the appli | |

# Appendix C Criteria for Identification of Markedly Abnormal Orthostatic Changes

| Davamatan | Cuitania | Changes |
|---|---|---|
| Parameter Orthostatic Hypotension | Criteria (Orthostatic Systolic Blood Pressure <-20 mi Orthostatic Diastolic Blood Pressure <-10 mi Heart Rate Increase >20 beats/min | n Hg OR<br>n Hg) AND |
| Note: Orthostatic measurement = stan | Heart Rate Increase >20 beats/min ding vital measurement - supine vital measurement. | 5 <del>6</del> // |
| | iect to the | |
| | and sulo, | |
| | SOULY S | |
| | cial use | |
| colfi | | |
| of nonre | | |
| egs. | | |
| x ale | | |
| O. T. | | |

# Appendix D Criteria for Markedly Abnormal Values for the 12-Lead ECG Parameters

| Parameter | Lower Criteria | Upper Criteria |
|---|---|---|
| Heart rate | <50 beats per minute | >120 beats per minute |
| PR | ≤80 milliseconds | ≥200 milliseconds |
| QT Interval | ≤300 milliseconds | ≥460 milliseconds |
| QTcB Interval | ≤300 milliseconds | ≥500 milliseconds OR |
| | | ≥30 milliseconds change from baseline <u>and</u><br>≥450 milliseconds |
| QTcF Interval | ≤300 milliseconds | ≥500 milliseconds OR |
| | | ≥30 milliseconds change from baseline <u>and</u> ≥450 milliseconds |
| QRS | ≤80 milliseconds | ≥180 milliseconds |

Property of Takeda. For non-commercial use only and supplements of the property of takeda.

# ELECTRONIC SIGNATURES

| Signed by | Meaning of Signature | Server Date (dd-MMM-yyyy HH:mm 'UTC') |
|---|---|---|
| PPD | Clinical Science Approval | 19-May-2017 19:47 UTC |
| | Statistical Approval | 19-May-2017 21:06 UTC |
| | Clinical Pharmacology Approval | 20-May 2017 00:58 UTC |
| | Pharmacovigilance Approval | 23-May-2017 19:50 UTC |
| | Clinical Approval | 25-May-2017 19:03 UTC |
| Property of Takeda. For non-comme | Rercial Use Only and sur | |